CLINICAL TRIAL: NCT04644848
Title: Diagnostic Accuracy of Preoperative Ultrasonographic Tattooing of Suspicious Axillary Lymph Nodes in Breast Cancer Patients With Clinically Negative Axilla. A Prospective Cohort Study.
Brief Title: Ultrasonographic Axillary Localization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of Surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R.20.11.1099
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasm
Keywords: sentinel lymph node biopsy; Axillary ultrasonography
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-sentinel node biopsy ultrasonographical tattooing (Experimental): Preoperative ultrasonographical tattooing of the suspicious lymph nodes. Sentinel Lymph Node Biopsy (SLNB),
  Interventions: Diagnostic Test: Ultrasonographical tattooing of suspicious axillary lymph nodes.; Procedure: Sentinel lymph node biopsy; Diagnostic Test: Histopathological examination of the axillary nodes; Procedure: Further axillary management

INTERVENTIONS:
Diagnostic Test: Ultrasonographical tattooing of suspicious axillary lymph nodes. — Patients with clinically negative axillae scheduled for sentinel lymph node biopsy (SLNB) will have axillary ultrasonographical imaging of the ipsilateral axilla with a high-frequency linear probe. Suspicious lymph nodes are identified according to any of the following criteria:
  * Round shape.
  * Cortical thickness > 3 mm
  * Eccentric cortical thickness.
  * Loss of hilum.
  For each patient, node dimensions and the presence of each of the above-mentioned criteria are recorded. Tattooing of all suspicious nodes is done using I ml of sterile liquid charcoal.
Procedure: Sentinel lymph node biopsy — Sentinel node biopsy is performed with peri-areolar subdermal injection of 3 ml methylene blue 5%. The lymphatics are tracked to the first blue lymph node. All blue, enlarged and /or tattooed nodes are separately biopsied and labelled as SLN and/or tattooed node.
Diagnostic Test: Histopathological examination of the axillary nodes — All tattooed nodes are excised and sent to frozen section examination; labelled tattoo node.
  All enlarged or blue stained nodes are excised and sent to frozen section examination; labelled sentinel node.
  All nodes are bisected and a single 5 um section examined. All frozen section examinations are followed by routine paraffin section examination.
Procedure: Further axillary management — Further axillary management is performed as per institutional guidelines. If SLNB is negative, no further surgery is required. Axillary lymph node dissection is performed if sentinel lymph node is positive or not identified. Management of positive SLNB as per the American College Of Surgeons' Oncology Group (ACOSOG) Z0011 protocol is not currently adopted on routine basis at the investigators' institution. In this study, patients with tattooed nodes with positive histopathological findings are offered full axillary dissection even if their sentinel nodes are negative.

SUMMARY:
Breast cancer is the most common cancer of women. Surgery for early breast cancer includes axillary lymph nodes staging. Axillary surgery may lead to intractable complications like permanent arm swelling. Axillary sentinel lymph node biopsy (SLNB) has been introduced to minimize the incidence of these complications. Several methods are routinely used for identification of the sentinel node during operation. Some of these methods necessitate facilities that are not universally available; specially in countries with limited resources. In its simplest form, SLNB using the methylene blue dye technique has an identification rate of 88-94%. If the sentinel node can not be identified, full axillary dissection may be required and the risk of arm swelling is increased. The objective of this study is to maximize the identification rate of the sentinel node thus avoiding the need for extensive axillary surgery. The investigators assumed that preoperative tattooing of the suspicious lymph node during ultrasonographical imaging may help the surgeon in localizing the sentinel lymph node. In this study, the sonographer will perform preoperative tattooing of the suspicious node. The surgeon will perform SLNB by the methylene blue dye. The sensitivity of ultrasonographical tattooing relative to SLNB will be calculated. The study will determine if the tattooing technique may localize additional nodes that are missed by the methylene blue.

DETAILED DESCRIPTION:
Introduction Axillary nodal staging is an integral part of breast cancer management. Sentinel lymph node biopsy (SLNB) has become a standard of care in patients with clinically negative axillae. Various methods have been investigated to decrease the false negative rate of SLNB. Ultrasonography is an established tool for preoperative axillary staging. The diagnostic accuracy of B-mode ultrasonographic criteria and of US-guided FNAC (Fine Needle Aspiration Cytology) has been described in the literature and its role in preoperative axillary staging has been emphasized.

Ultrasonographic aspiration of suspicious axillary nodes are widely used to identify axillary metastases and obviate the need for SLNB. Previous studies retrospectively examined the concordance of ultrasonographic identification of suspicious lymph nodes with subsequent SLNB results. However, ultrasonographic axillary staging have not been prospectively compared to SLNB. In addition, concomitant ultrasonographic and SLNB are thought to increase the overall accuracy of axillary staging.

In this study, the investigators will perform preoperative ultrasonographic axillary evaluation and tattooing of suspicious lymph nodes followed by SLNB with methylene blue technique. Head-to-head and node-to-node comparison of ultrasonographic and surgical staging will be conducted.

Specific aims

1. Determination of the diagnostic accuracy of preoperative ultrasonic guided tattooing of suspicious axillary lymph nodes.
2. Determination of node-to-node concordance of ultrasonographic tattooing relative to blue dye SLNB.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven invasive breast adenocarcinoma.
* Clinically non palpable axillary lymph nodes.
* T0-3, N0, M0
* Scheduled for definitive surgery.

Exclusion Criteria:

* Patient unwilling to participate.
* Contraindication to methylene blue technique: hypersensitivity, pregnancy.
* T4 primary tumor.
* Previous axillary surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ultrasonographical tattooing | at the date of surgery.
  The ratio of the tattooed lymph nodes (that are positive by histopathological examination) to the sentinel lymph nodes (that are positive by histopathological examination).
Identification benefit of the ultrasonographical tattooing. | at the date of surgery.
  The ratio of the cases with successfully tattooed nodes and non identified sentinel node to the total number of analyzed cases.

OTHER OUTCOMES:
Negative predictive value of ultrasonographical tattooing. | at the date of surgery.
  The ratio of tattooed nodes (that are negative by histopathological examination) to the sentinel lymph nodes (that are negative by histopathological examination).
Concordance of ultrasonographical tattooing with sentinel lymph nodes. | at the date of surgery.
  The ratio of cases that have similar histopathological examination results (of both tattooed and sentinel nodes) to the total number of analyzed cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim WH, Kim HJ, Jung JH, Park HY, Lee J, Kim WW, Park JY, Cheon H, Lee SM, Cho SH, Shin KM, Kim GC. Ultrasound-Guided Fine-Needle Aspiration of Non-palpable and Suspicious Axillary Lymph Nodes with Subsequent Removal after Tattooing: False-Negative Results and Concordance with Sentinel Lymph Nodes. Ultrasound Med Biol. 2017 Nov;43(11):2576-2581. doi: 10.1016/j.ultrasmedbio.2017.07.011. Epub 2017 Aug 19. PMID 28830644
- [Background] Li J, Chen X, Qi M, Li Y. Sentinel lymph node biopsy mapped with methylene blue dye alone in patients with breast cancer: A systematic review and meta-analysis. PLoS One. 2018 Sep 20;13(9):e0204364. doi: 10.1371/journal.pone.0204364. eCollection 2018. PMID 30235340